CLINICAL TRIAL: NCT05631990
Title: A Randomized, Double-Blind, Parallel, Multi-Center, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of AD-209 in Patients With Essential Hypertension
Brief Title: A Study to Evaluate the Efficacy and Safety of AD-209
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-209P2-02
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Hypertension, Essential
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental 1 (Experimental): AD-209, AD-209-1 placebo
  Interventions: Drug: AD-209; Drug: AD-209-1 placebo
- Experimental 2 (Experimental): AD-209-1A, AD-209 placebo
  Interventions: Drug: AD-209-1A; Drug: AD-209 placebo
- Experimental 3 (Experimental): AD-209-1B, AD-209 placebo
  Interventions: Drug: AD-209-1B; Drug: AD-209 placebo
- Experimental 4 (Experimental): AD-209-1C, AD-209 placebo
  Interventions: Drug: AD-209-1C; Drug: AD-209 placebo

INTERVENTIONS:
Drug: AD-209 — PO, Once daily(QD), 8weeks
  Arms: Experimental 1
Drug: AD-209-1A — PO, Once daily(QD), 8weeks
  Arms: Experimental 2
Drug: AD-209-1B — PO, Once daily(QD), 8weeks
  Arms: Experimental 3
Drug: AD-209-1C — PO, Once daily(QD), 8weeks
  Arms: Experimental 4
Drug: AD-209 placebo — PO, Once daily(QD), 8weeks
  Arms: Experimental 2; Experimental 3; Experimental 4
Drug: AD-209-1 placebo — PO, Once daily(QD), 8weeks
  Arms: Experimental 1

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of AD-209

DETAILED DESCRIPTION:
Condition or disease : hypertension Intervention/treatment Drug : AD-209 Drug : AD-209-1A Drug : AD-209-1B Drug : AD-209-1C Drug : AD-209 Placebo Drug : AD-209-1 Placebo Phase : Phase 2

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Other inclusions applied

Exclusion Criteria:

* orthostatic hypotension with symptom
* Other exclusions applied

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Change rate of MSSBP | Baseline, Week 8
  Change from baseline in mean sitting systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Chang Gyu Park, M.D., Ph.D, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No